CLINICAL TRIAL: NCT06652165
Title: A Single-center, Randomized Controlled Clinical Study of Zanubrutinib Combined With Carmustine, Etoposide, Cytarabine, and Melphalan (BEAM) as a Preconditioning Regimen for ASCT in Relapsed and Refractory DLBCL
Brief Title: Zanubrutinib Combined With BEAM for ASCT in Relapsed and Refractory DLBCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASCT-003
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-08

CONDITIONS: DLBCL

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- zanubrutinib combined with BEAM (Experimental): zanubrutinib combined with camustine, etoposide, cytarabine, and mafaran (BEAM)
  Interventions: Drug: zanubrutinib combined with BEAM
- BEAM (Active Comparator): camustine, etoposide, cytarabine, and mafaran (BEAM)
  Interventions: Drug: BEAM

INTERVENTIONS:
Drug: zanubrutinib combined with BEAM — zanubrutinib：160mg oral bid D-8-D-2 camustine: 300mg/m2 vgtt qd D-8 etoposide: 100mg/m2/d vgtt q12h D-7-D-4 cytarabine: 200mg/m2/d vgtt q12h D-7-D-4 melphalan: 140mg/m2 vgtt qd D3-D-2
  Arms: zanubrutinib combined with BEAM
Drug: BEAM — camustine: 300mg/m2 vgtt qd D-8 etoposide: 100mg/m2/d vgtt q12h D-7-D-4 cytarabine: 200mg/m2/d vgtt q12h D-7-D-4 melphalan: 140mg/m2 vgtt qd D3-D-2
  Arms: BEAM

SUMMARY:
This trial is a prospective, single-center, randomized controlled clinical research. The intention is to evaluate the efficacy and safety of zanubrutinib combined with BEAM as a pretreatment regimen for ASCT in relapsed and refractory DLBCL patients through prospective clinical studies.

DETAILED DESCRIPTION:
This trial includes 66 patients with recurrent or refractory DLBCL, who will be randomly divided into a 1:1 combination of zanubrutinib and BEAM regimen pretreatment (experimental group) or a standard BEAM regimen pretreatment (control group), and then undergo ASCT treatment. The entire trial includes a screening period (before the start of autologous stem cell transplantation pretreatment), a treatment period (-8 days to -2 days, a total of 7 days), and a follow-up period (2 years after autologous stem cell transplantation)

ELIGIBILITY:
Inclusion Criteria:

1. According to world Health Organization (WHO) classification of disease, diffuse large B-cell lymphoma was confirmed by histology, CR or PR after second-line and above treatment;
2. 18≤ age ≤65 years old, male or female;
3. ECOG score 0-2;
4. No serious organic lesions in the main organs, meeting the requirements of the following laboratory examination indicators (conducted within 7 days before treatment) :

   1. White blood cell count ≥3.0×109/L, absolute neutrophil count ≥1.5×109/L, Hemoglobin ≥90g/L, platelet ≥75×109/L;
   2. Total bilirubin ≤1.5× upper normal value (ULN);
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5× ULN; Bilirubin ≤1.5× ULN
   4. Creatinine clearance was 44-133 mmol/L;
5. No cardiac dysfunction;
6. Life expectancy over 3 months;
7. The subject or his/her legal representative must provide written informed consent prior to conducting a special study examination or procedure.

Exclusion Criteria:

1. Previously received autologous hematopoietic stem cell transplantation;
2. Suffering from serious complications or severe infection;
3. Previous treatment with selinexor;
4. Central nervous system lymphoma was excluded;
5. A history of other malignant tumors within 5 years, excluding early tumors treated for curative purposes;
6. Patients with uncontrolled cardiovascular and cerebrovascular diseases, coagulation disorders, connective tissue diseases, serious infectious diseases, etc.;
7. HBsAg, HCV or HIV positive. Positive HBV and HCV serology is allowed, but DNA/RNA testing must be negative;
8. Left ventricular ejection fraction ≦ 50%;
9. Laboratory test value during screening;

   ① Neutrophils <1.5×109/L; Platelet <75×109/L;

   ② Bilirubin was 1.5 times higher than the normal upper limit, transaminase was 2.5 times higher than the normal upper limit;

   ③ The creatinine level is higher than 1.5 times the upper limit of normal value;
10. Other concurrent and uncontrolled medical conditions considered by the investigator would affect the patient's participation in the study;
11. Psychiatric patients or other patients known or suspected to be unable to fully comply with the study protocol;
12. Pregnant or lactating women;
13. The researcher judged that the patients were not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Baseline up to data cut-off (up to approxiamately 2 years)
  Progression-free survival was defined as the time from the data of ASCT until the date of the first documented day of disease progression or relapse, using Lugano criteria, or death from an cause, whichever occured first.

SECONDARY OUTCOMES:
Overall survival | Baseline up to data cut-off (up to approxiamately 2 years)
  Overall survival was defined as the time from the date of ASCT to the date of death from any cause
Complete remission rate | 3 months after the transplantation
  Percentage of participants with complete response was determined on 2014 Lugano criteria
The time of hematopoietic reconstruction | 2 months after the transplantation
  The first day of neutrophils ≥0.5*109/L for 3 consecutive days was the time of successful implantation of granulocytes. Platelet ≥20.0*109/L for 7 consecutive days and the first day after platelet infusion was considered as the successful time of megakaryocytes implantation
Transplantation-related adverse reactions | Baseline up to data cut-off (up to approxiamately 4 years)
  Transplantation-related adverse reactions are any untoward medical occurrence in a participant which is related to ASCT.

IPD SHARING:
Plan to Share IPD: No